CLINICAL TRIAL: NCT00964574
Title: Multicentre, Open, Non-randomised Controlled Phase IV Clinical Trial of Efficacy and Safety for Insulin Glulisine Injected Subcutaneously in Patients With Type 1 Diabetes Mellitus Using Also Insulin Glargine
Brief Title: Test of the Efficacy and Safety of Insulin Glulisine Injected Subcutaneously in Patients With Type 1 Diabetes Mellitus
Acronym: PORTAL 1
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APIDR_L_02483
Record Dates: First submitted 2009-08-24; First posted 2009-08-25 (Estimated); Last update posted 2012-07-17 (Estimated); Status verified 2012-07

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — insulin glulisine; Insulin Glargine

ARMS (1):
- APIDRA + LANTUS basal (Experimental): The 2 first weeks, patients will receive subcutaneous injection of Insulin Glulisine and Insulin Glargine once daily in hospital. The rest of the treatement is to be take at home until week 12
  Interventions: Drug: INSULIN GLULISINE (HMR1964); Drug: INSULIN GLARGINE

INTERVENTIONS:
Drug: INSULIN GLULISINE (HMR1964) — Pharmaceutical form:
  APIDRA 100U/ml flacon for the titration period in the hospital APIDRA 100U/ml solution for injection in cartridge in OptiSet
  Route of administration:
  3-4 subcutaneous injections per day
Drug: INSULIN GLARGINE — Pharmaceutical form:
  LANTUS 100U/ml solution for injection in cartridge
  Route of administration:
  Once daily subcutaneous injection in the evening

SUMMARY:
Primary Objective:

To evaluate the efficacy and the safety of insulin glulisine in type I Diabetes Melittus (DM) patients

Secondary Objective:

To evaluate the insulin glulisine doses To assess the patient satisfaction

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 1 diabetes mellitus who need insulin basal+ bolus regimen
* 6.5 <=HbA1c <= 11% at visit 1
* BMI <35 kg/m²
* Provision of signed and dated informed consent prior to any study procedures
* Ability and willingness to complete study diaries and questionnaires
* Demonstrated ability to use the self-glucose-monitoring device, and to self-inject insulin
* A negative pregnancy test for all females of childbearing potential.

Exclusion criteria:

* Hypersensitivity to insulin Glulisine, insulin Glargine or one of their excipients
* Pregnant women
* Active proliferative diabetic retinopathy
* Impaired hepatic or renal function

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2009-07; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Mean change in Glycosylated haemoglobin (HbA1c) | Week 12

SECONDARY OUTCOMES:
Mean Glycosylated haemoglobin (HbA1c) | Week 12
Mean Fasting Blood Glucose and mean Post Prandial Glycemia | Week 12
Number of documented symptomatic hypoglycaemic episodes | From week 0 to week 12
Mean dose and mean dose change of insulin glulisine, basal glulisine and total insulin from baseline | week 12
Mean change of Fasting Blood Glucose and Post Prandial Glycemia | From week 0 to week 12

CONTACTS AND LOCATIONS:
Overall Officials: Natallia Zhyhaila, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis Administrative Office, Minsk, Belarus